CLINICAL TRIAL: NCT07391410
Title: The International Bone Metastasis Registry
Brief Title: Registry for Bone Metastases
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-175
Record Dates: First submitted 2026-01-23; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Bone Metastases
Keywords: 23-175

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bone Metastases

SUMMARY:
The purpose of this study is to learn more about symptomatic bone metastases. This study is an international patient registry of people with symptomatic bone metastases. A patient registry is a database - a collection of health information - about a group of people, and it is usually focused on a specific diagnosis or condition.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥22 years
* Biopsy-proven or clinically obvious metastatic bone disease
* Symptomatic bone lesion requiring intervention
* This includes but is not limited to radiotherapy, cryotherapy, radiofrequency ablation, operative fixation, prosthetic replacement, amputation, or any combination of the above

Exclusion Criteria:

* Age <22 years

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There is also a retrospective component to this study, in which we will review data on patients going back to 2015; we will analyze data from any patients who died with symptomatic metastatic bone disease for possible inclusion in the IBMR. Living patients will be prospectively enrolled into the trial.
  For the retrospective component, only deceased patients (500) will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Forsberg, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/